CLINICAL TRIAL: NCT04307524
Title: Laparoscopic Repair Of Cesarean Scar Niche: Randomized Controlled Trial.
Brief Title: Laparoscopic Repair of Cesarean Scar Niche
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Mahmoud Ismail Abdel Rahman Kotb, Specialist & Assistant Lecturer of obstetrics and gynecology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: cesarean scar niche
Record Dates: First submitted 2020-02-21; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Cesarean Section Complications
Keywords: cesarean scar niche

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: computer-generated sequence
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- laparoscopic repair (Experimental): suture repair of cesarean scar niche using laparoscopy
  Interventions: Procedure: laparoscopic repair
- medical treatment (Active Comparator): conservative management
  Interventions: Drug: medical treatment in the form of combined hormonal contraception

INTERVENTIONS:
Procedure: laparoscopic repair — laparoscopic suture repair of cesarean scar niche
  Arms: laparoscopic repair
Drug: medical treatment in the form of combined hormonal contraception — patient will receive for three months daily without interruption, no pill-free interval drug names is "Genera" BAYERhealthcare
  Arms: medical treatment

SUMMARY:
Evaluation of laparoscopy repair of cesarean scar niche in resolution of symptoms related to niche as compared to expectant management.

DETAILED DESCRIPTION:
Recently, The percentage of Cesarean section (CS) deliveries has dramatically increased in most countries. The presence of a niche at the site of a CS scar has been observed. A niche is mainly a sonographic finding defined as a triangular anechoic area at site of incision. ( Mascarello et al, 2017) Alternative terms for a niche are Cesarean scar defect (Wang et al, 2009), deficient Cesarean scar (Ofili-Yebovi et al, 2008), diverticulum (Surapaneni et al, 2008), pouch (Fabres el al, 2003) and isthmocele. (bogres el al, 2010) As not all women with previous CS develop a niche, it is a matter of interest to identify the risk factors that may predict their development. (Sholapurkar , 2018) Possible causes of this condition may be surgery or patient related. Surgery related factors as low cervical incision, incomplete closure of the uterus (decidual sparing) and inadequate hemostasis. Patient related factors may be attributed to infection. ( Vervoort et al, 2015) Cesarean scar niche may be asymptomatic or may cause a number of obstetrical and gynecological problems (cesarean scar syndrome) . ( Vervoort et al,2015b) Obstetrical complications of the niche are cesarean scar ectopic pregnancy, placenta previa and morbidly adherent placenta, cesarean scar dehiscence following incomplete abortion secondary to uterotonic drugs, Scar dehiscence and tender scar even scar rupture (Tanimura el al, 2015) Gynecological symptoms of the niche are postmenstrual spotting, Intermenstrual bleeding, Dysmenorrheal, Dysparunia and secondary infertility. (Tanimura el al, 2015) Various methods to detect and measure a niche have been described. The majority of papers have evaluated the niche with the use of transvaginal sonography (TVS) (Vaate et al, 2011), and contrast-enhanced sonohysterography (SHG) (Bij de Vaate et al, 2011), but a minority have used hysteroscopy (El-Mazny et al, 2011) or hysterosalpingography. (Surapaneni and Silberzweig, 2008 ) At present there is no consensus regarding the gold standard for the detection and measurement of a niche. (Vaate et al, 2014) Symptomatic cesarean scar niche (cesarean scar syndrome) can be managed conservatively using combined oral contraceptive pills especially in women not seeking fertility, or it can be treated using minimal invasive surgery as hysteroscopic resection (vervoot et al,2017) , laparoscopic repair (ma et al,2017) or vaginal repair (Yao, 2014) In this study we will evaluate laparoscopic management of cesarean scar niche

ELIGIBILITY:
Inclusion Criteria:

1. History of cesarean section.
2. Postmenstrual and/or intermenstrual spotting.
3. Cesarean scar niche of at least 2 mm in depth diagnosed by saline infusion sonography

Exclusion Criteria:

1. pregnancy
2. Uterine anomalies
3. Hysterotomy.
4. history Placenta previa and MAP
5. Upper segment incision, Vertical uterine incision
6. submucosal fibroids
7. adenomyosis.
8. History atypical endometrial cells, cervical dysplasia,
9. cervical or pelvic infection.
10. Irregular cycle.
11. lactation amenorrhea.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-03-15 (Estimated); Primary Completion 2021-03-15 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
post-menstrual spotting | 6 month after intervention
  number of days of post-menstrual spotting "spotting or bleeding after 8 days of menstruation whatever the amount

SECONDARY OUTCOMES:
menstrual related pain | 6 month after intervention
  degree of menstrual related pain as descriped by the patient on Visual Analogue Scale of pain from 1 to 10
infertility | 6 month after intervention
  failure of conception despite regular sexual intercourse within 6 months from intervention or stopping gynera

IPD SHARING:
Plan to Share IPD: No